CLINICAL TRIAL: NCT03356730
Title: Effect of Vitamin D Replacement on Bone Healing in Mini-dental Implants: a Randomized Clinical Trial
Brief Title: Effect of Vitamin D Replacement on Bone Healing in Mini-dental Implants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade de Passo Fundo (Other)
Responsible Party: Principal Investigator, Isadora Rinaldi, Master Student, Universidade de Passo Fundo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UPassoFundo
Record Dates: First submitted 2017-08-17; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Deficiency, Vitamin D
Keywords: Implants; Vitamin D; Osseointegration; Histomorphometric
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: This is a clinical research study, characterized by a randomized, double-blind, placebo-controlled trial.
Who Masked: Participant, Investigator
Masking Description: Masking for placebo or vitamin D use
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm vitamin D (Experimental): Vitamin D 5.000 IU a day for 2 months (10 drops after lunch)
  Interventions: Drug: Vitamin D
- Arm placebo (Placebo Comparator): Placebo for 2 months (10 drops after lunch)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin D — Only patients with vitamin D deficiency / deficiency will be included in the study. Randomly, they will be divided into two groups. This group will receive vitamin D supplementation.
  Vitamin D3 - cholecalciferol, oral suspension in drops, will be prescribed as follows:
  • 5,000 IU / day - 10 drops per day for two months.
  Arms: Arm vitamin D
Other: Placebo — Only patients with vitamin D deficiency / deficiency will be included in the study. Randomly, they will be divided into two groups. This control group will receive placebo.
  Placebo (olive oil mint flavor), oral suspension in drops, will be prescribed as follows:
  • 10 drops per day for two months.
  Arms: Arm placebo

SUMMARY:
1. Title
2. Executive team
3. Research line
4. Summary
5. Research problem
6. Justification
7. Literature review
8. Objectives
9. Materials and methods
10. Dissemination of knowledge generated
11. Schedule of activities
12. Budget
13. References
14. Annexes

DETAILED DESCRIPTION:
This is a clinical research study, characterized by a randomized, double-blind, placebo-controlled clinical trial. Background: Vitamin D replacement could aid in the osseointegration of dental implants. Objective: to evaluate the effect of vitamin D replacement on osseointegration of dental implants in humans. Materials and methods: Twenty individuals with hypovitaminosis D underwent dental miniimplants and randomized to two equal groups for treatment with vitamin D (5000 IU / day) or placebo for 2 months. After two months, the miniimplants will be removed and prepared for histomorphometric analysis, which will evaluate bone implant contact in percentage. Testing the hypothesis that the contact between bone and implant and the bone density in the threaded area in the test group is higher than in the control group. Test t will be used to compare the differences between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes;
* No medical, temporary or intra-oral contraindications;
* Good general health;
* Need of implant in the maxilla in the posterior region (with a minimum of 5 mm of bone height visualized radiographically) or in mandible in posterior region;
* With vitamin D deficiency / deficiency (considering serum level of ≥ 15 ng / ml at ≤ 25 ng / ml).

Exclusion Criteria:

* Medical, temporary or intrabuccal contraindications;
* Smokers;
* Use of corticoid;
* Post-operative of bariatric surgery;
* Bone height less than 5mm;
* Need for maxillary sinus lift;
* Vitamin supplementation D.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11-19 (Actual); Primary Completion 2017-12-30 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of bone implant contact | 2 months
  Histomorphometry will be used as a method of analysis. It will evaluate the initial stage of osseointegration in the two groups, relating it to insufficiency / deficiency and sufficiency of vitamin D. The percentage of bone implant contact, defined as the amount of mineralized bone in direct contact with the surface of the miniimplant, will be evaluated.

SECONDARY OUTCOMES:
Serum levels of vitamin D (ng/ml) | 2 months
  The 25-hydroxyvitamin D test is a common blood test and is the best way to monitor vitamin D levels. The test can determine if the person's blood has deficiency or excessive vitamin D. The method used to evaluate the blood test is chemiluminescent immunoassay technology (CLIA).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Salete Sandini Linden, Study Director — Universidade de Passo Fundo
Locations (1):
- Isadora Rinaldi, Rondinha, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The individual participants data (IPD) will be available in the dental records including complementary exams, allowing the access of other researchers during the research.